CLINICAL TRIAL: NCT05162664
Title: Presence of Signs of Central Sensitization in Episodic and Chronic Migraine - a Cross Sectional Study
Brief Title: Presence of Signs of Central Sensitization in Episodic and Chronic Migraine
Acronym: CENSENMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: BC-08688
Record Dates: First submitted 2021-09-27; First posted 2021-12-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Central Sensitisation; Migraine
Keywords: Migraine; Headache; PPT; CPM; Pain
MeSH Terms: conditions — Migraine Disorders; Headache; Pain | interventions — Pain Threshold; Postsynaptic Potential Summation

STUDY DESIGN:
Intervention Model Description: Cross-sectional study, in which patients with migraine are gender- and age matched to healthy controls, and undergo a pain protocol.
Who Masked: Outcomes Assessor
Masking Description: In total, three investigators are involved. One is in charge for the screening process, and is not blinded for the status of the participants. The second investigator, i.e. the outcome assessor, is blinded for the status of the participants, and performs the clinical assessments (NOT the questionnaires). A third senior researcher is supervising the process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (Other): Healthy controls
  Interventions: Other: Pressure pain thresholds; Other: Thermal detection and pain thresholds; Other: Temporal summation; Other: Conditioned pain modulation
- Patients with migraine (Other)
  Interventions: Other: Pressure pain thresholds; Other: Thermal detection and pain thresholds; Other: Temporal summation; Other: Conditioned pain modulation

INTERVENTIONS:
Other: Pressure pain thresholds — PPT will be performed firstly at the anterior tibial muscle halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly (13) and secondly at the middle of the temporalis muscle (12), using a digital algometer (Wagner FPX 50) with a 1 cm2 rubber tip. The pressure algometer will apply a perpendicular increasing pressure (1kg/s) at the different test locations until the participant reports the first feeling of pain. The PPT of 4 series of ascending stimulus intensities, with an inter-stimulus interval (ISI) of 20sec between the different stimuli and an ISI of 60sec between the 2 locations, will be measured. The first stimulus is a familiarization stimulus. Afterwards the mean of the 3 subsequent stimuli will be calculated.
Other: Thermal detection and pain thresholds — The thermal tests will be performed unilateral at tibial anterior, thenar and the forehead, using a TSA-2 (Neuro Sensory Analyzer, MEDOC). At first cold and heat detection thresholds will be measured. The patient will be asked to indicate when they feel a change in temperature. Afterwards the patient will be asked to indicate when the stimulus becomes painful to determine the cold and heat pain thresholds. The thresholds of 4 series of stimuli will be measured. The first stimulus is a familiarization stimulus. Afterwards the mean of the 3 subsequent stimuli will be calculated for every location. The subject will push a button when the thresholds are reached. The baseline temperature will be 32°C and the stimuli will increase with 1°C/s (14).
Other: Temporal summation — The temporal summation will be assessed at the thenar eminence (19,20) using a ramp and hold protocol with the TSA-2 (Neuro Sensory Analyzer, MEDOC). Heat stimuli will be applied for a duration of 15sec. The stimulus temperature will increase from a baseline temperature of 35°C for 9sec at a sensitivity-adjusted rate of about 1,5°C/s until the HTP 5/10 of the thenar is reached. Afterwards the temperature will remain steady for the next 6 seconds. The maximal pain rating should be 50 ± 10 NRS. Subjects rate the pain intensity at the end of the ramp (9sec) and at the end of the hold procedure (15sec) using the NRS. Afterwards the ramp and hold aftersensations are measured. The subjects have to rate the pain intensity every 5sec for 30sec after the termination of the heat stimulus.
Other: Conditioned pain modulation — CPM will be assessed by comparing heat pain thresholds and pressure pain thresholds before and after giving a conditioning stimulus at a pain free distant zone by using a second thermode of the TSA-2 (17). The conditioning stimulus (HPT 4/10 (18) at the TA) will be applied for 120 seconds. The first test stimulus will be applied at the forehead 30 seconds after the start of the conditioning stimulus (17). The HPT will be measured twice with an ISI of 20 seconds. Immediately after the end of the application of the conditioning stimulus (120 seconds), the HPT at the forehead will be measured again twice, with an ISI of 20 seconds. Afterwards, there will be 10 minutes of rest to avoid bias.

SUMMARY:
Nowadays migraine is conceptualized as a continuum, with at the one hand episodic migraine (EM) and at the other hand chronic migraine (CM) (1). The general aim of the study is to determine where exactly in this continuum central sensitization (CS) appears.

Recent studies support the presence of CS in migraine patients (2,3), but controversial evidence exists about where in the continuum exactly CS appears. Some studies determined no differences in sings of CS between EM and CM (4,5), whether other research indicate a clear difference between EM and CM (6-8). However a significant difference in CS parameters could be determined between a patient group (EM or CM) and a healthy control group (3,4,8). In addition, CS appears to be present during the migraine attack (2). In this research, the presence of signs of CS will be determined in between headache phases.

The primary outcome measure is identification of CS by PPT, QST, TS, CPM and CSI. Secondary outcome measures are the outcome of the MIDAS, HADS and EUROLIGHT.

DETAILED DESCRIPTION:
For objectifying central sensitization, both self-reported and psychophysiological measures of allodynia and hyperalgesia will be used. These symptoms are considered to be signs of central sensitization, especially when present at distant pain-free areas (9).

Therefore, 100 patients with migraine (50 EM, 50 CM) and 50 healthy controls will be recruited. The patients should meet the following inclusion criteria: 1) diagnosis of migraine headache based on the criteria of ICDH-3 and verified by a medical doctor, 2) not being pregnant or have given birth in the preceding year, 3) adults between the age of 18 years and 65 years. Exclusion criteria are: 1) any other diagnosis of headache or mixed form, 2) any structural neurological syndrome, 3) any neurological brain event in the past, 4) surgery at the head, neck or shoulder the last 3 years.

As thermal testing might be followed by a mechanical hyperalgesia (10), this protocol will start with evaluating the mechanical sensitivity and afterwards the thermal sensitivity. The mechanical sensitivity will be determined by measuring PPT (A). A standardized and reliable QST protocol (B), including detection and sensitivity to warmth and cold, will be used (11). The temporal summation (C) will be used to asses endogenous pain facilitating pathways and conditioned pain modulation (CPM) (D) will be used to assess the endogenous pain inhibitory pathways. In addition questionnaires (E) will be conducted. The patients will be tested unilateral at the painful side and interictally.

Pressure pain thresholds PPT will be performed firstly at the anterior tibial muscle halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly (13) and secondly at the middle of the temporalis muscle (12), using a digital algometer (Wagner FPX 50) with a 1 cm2 rubber tip. The pressure algometer will apply a perpendicular increasing pressure (1kg/s) at the different test locations until the participant reports the first feeling of pain. The PPT of 4 series of ascending stimulus intensities, with an inter-stimulus interval (ISI) of 20sec between the different stimuli and an ISI of 60sec between the 2 locations, will be measured. The first stimulus is a familiarization stimulus. Afterwards the mean of the 3 subsequent stimuli will be calculated.

Thermal detection and pain thresholds The thermal tests will be performed unilateral at tibial anterior, thenar and the forehead, using a TSA-2 (Neuro Sensory Analyzer, MEDOC). At first cold and heat detection thresholds will be measured. The patient will be asked to indicate when they feel a change in temperature. Afterwards the patient will be asked to indicate when the stimulus becomes painful to determine the cold and heat pain thresholds. The thresholds of 4 series of stimuli will be measured. The first stimulus is a familiarization stimulus. Afterwards the mean of the 3 subsequent stimuli will be calculated for every location. The subject will push a button when the thresholds are reached. The baseline temperature will be 32°C and the stimuli will increase with 1°C/s (14). The contact area of the thermode will be 16mm x 16mm. The cut-off temperature for heat is 53°C and for cold 0°C. The ISI will be 20 seconds on one location, and 1min between different locations. After measuring a thermal detection threshold, the temperature will go back to baseline with 1°C/s and after a thermal pain threshold measurement with 5°C/s.

The tibial anterior muscle will be measured halfway between the most superior attachment to the tibia and its tendon in the upper one third of the muscle belly (13).

The hand will be measured at the thenar eminence overlying the abductor pollicis brevis muscle (15).

The forehead will be measured in the supra-orbital area, within the territory of the ophthalmic division of the trigeminal nerve (14).

Temporal summation (19) The temporal summation will be assessed at the thenar eminence (19,20) using a ramp and hold protocol with the TSA-2 (Neuro Sensory Analyzer, MEDOC). Heat stimuli will be applied for a duration of 15sec. The stimulus temperature will increase from a baseline temperature of 35°C for 9sec at a sensitivity-adjusted rate of about 1,5°C/s until the HTP 5/10 of the thenar is reached. Afterwards the temperature will remain steady for the next 6 seconds. The maximal pain rating should be 50 ± 10 NRS. Subjects rate the pain intensity at the end of the ramp (9sec) and at the end of the hold procedure (15sec) using the NRS. Afterwards the ramp and hold aftersensations are measured. The subjects have to rate the pain intensity every 5sec for 30sec after the termination of the heat stimulus.

Conditioned pain modulation The CPM effect appears to reduce when CS is present (16). CPM will be assessed by comparing heat pain thresholds and pressure pain thresholds before and after giving a conditioning stimulus at a pain free distant zone by using a second thermode of the TSA-2 (17). The conditioning stimulus (HPT 4/10 (18) at the TA) will be applied for 120 seconds. The first test stimulus will be applied at the forehead 30 seconds after the start of the conditioning stimulus (17). The HPT will be measured twice with an ISI of 20 seconds. Immediately after the end of the application of the conditioning stimulus (120 seconds), the HPT at the forehead will be measured again twice, with an ISI of 20 seconds. Afterwards, there will be 10 minutes of rest to avoid bias. The conditioning stimulus will be applied for 120 seconds another time. The second test stimulus (PPT) will be applied twice at the forehead 30 seconds after the start of the conditioning stimulus, with an ISI of 20 seconds, and twice immediately after the end of the conditioning stimulus (120 seconds), with an ISI of 20 seconds. The HPT and PPT of the test stimulus is calculated as the mean of 2 consecutive trials, for the parallel and sequential protocol separate.

The effect of CPM will be calculated as (TSpostCS - TSpreCS) whereby a negative value corresponds with an inhibition and a positive value with a facilitation (18).

Test stimulus: HPT forehead and PPT forehead Conditioning stimulus: HPT 4/10 TA

Questionnaires Demographic questionnaire A questionnaire including questions concerning age, sex, history, socio-economic factors, and headache specific factors will be conducted. Within the headache specific factors, attention will be paid to the headache phase the patient is in and whether or not the headache is associated with an aura.

Clinical symptoms questionnaire A questionnaire including questions concerning clinical symptoms that indicate the presence of central sensitization (21,22).

Migraine Disability Assessment Questionnaire The MIDAS is a self-reported questionnaire about the impact of migraine headache on the daily functioning (23).

Central Sensitization Inventory The CSI is a self-reported questionnaire that assesses symptoms indicative of central sensitization. The CSI has proven psychometric strength (24,25).

Hospital Anxiety and Depression Scale The HADS will give an overview of present symptoms of anxiety and depression, without involving the physical complaints, by focusing on feelings the last period. This questionnaire has proven to be a reliable and valid assessment tool (26,27).

EUROLIGHT questionnaire The EUROLIGHT questionnaire is a self-reported questionnaire to assess the burden of primary headache disorders on those affected by them, including headache characteristics, associated disability, co-morbidities, disease management and quality of life. The questionnaire has proven psychometric strength (28).

Procedure Each subject participated, during the interictal phase, in 1 experimental session of 1h30. A baseline questionnaire was send 3 days before the testing. If a migraine attack occurred within 3 days before or after the testing day, the researcher was contacted and another testing moment was scheduled. The clinical symptoms questionnaire was administered at the day of the testing, by the researcher. Afterwards the subject was side lying position. The PPT at TA was measured by placing the algometer perpendicular at the TA. For the PPT forehead, the patient was placed in supine position. The thermal detection and pain thresholds, temporal summation and conditioned pain modulation were measearud in supine position. The patient could not see the screen of the computer. The researcher was blinded for the PPT measurement as this could bias the results.

ELIGIBILITY:
The patients should meet the following inclusion criteria:

1. diagnosis of migraine headache based on the criteria of ICDH-3 and verified by a medical doctor,
2. not being pregnant or have given birth in the preceding year,
3. adults between the age of 18 years and 65 years.

Exclusion criteria are:

1. any other diagnosis of headache or mixed form,
2. any structural neurological syndrome, 3) any neurological brain event in the past,

4) surgery at the head, neck or shoulder the last 3 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Extend of central sensitization by quantitative sensory testing (QST) in °C. | at baseline
  The primary outcome will include heat detection treshold and heat pain treshold.
Extend of Central sensitization by central sensitization inventory (CSI) as a scale | at baseline
  The primary outcome will include the score of each participant on the CSI questionnaire.

SECONDARY OUTCOMES:
Extend of Disability measured by the MIDAS questionnaire. | at baseline
  The score of the MIDAS questionnaire for each participant will be recorded.
Extend of Anxiety and depression measured by the HADS questionnaire. | at baseline
  The score of the HADS questionnaire for each participant will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No